CLINICAL TRIAL: NCT02682095
Title: Possibilities for Patients With Elevated Blood Pressure to Achieve Blood Pressure Control Without Affecting Quality of Life (the PEQ Study)
Brief Title: To Achieve Blood Pressure Control With Retained Quality of Life
Status: Terminated | Type: Observational
Why Stopped: Only part three, the individual interviews, has been carried out. We have not been able to get funding to complete the rest of the study.
Sponsor: Eva Drevenhorn (Other)
Responsible Party: Sponsor-Investigator, Eva Drevenhorn, Senior Lecturer, Lund University
Organization: Lund University (Other)
Other Study IDs: The PEQ-study
Record Dates: First submitted 2016-02-08; First posted 2016-02-15 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Hypertension; Patient Compliance
Keywords: Hypertension; Blood Pressure Control; Adherence; Mixed Methods
MeSH Terms: conditions — Hypertension; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Patients: achieved BP control: Patients who have achieved blood pressure control (≤140/90 mmHg)
- Patients: not achieved BP control: Patients who have not achieved blood pressure control (>140/90 mmHg)
- Individual interviews: Hypertensive patients who have considered changing lifestyle regarding one or more of the areas of tobacco, alcohol, diet, physical activity or stress.
- Focus-group interviews: Hypertensive patients

SUMMARY:
The purpose of the study is to get an understanding about what problems patients with hypertension are facing, how they manage these challenges, how they feel and what requirements they believe are important to have in their treatment. These factors will later act as a foundation and incentive for designing an intervention that may result in more patients achieving blood pressure control with maintained quality of life.

DETAILED DESCRIPTION:
This is a Swedish observational mixed-methods study to get an understanding about what problems patients with hypertension are facing. The information will act as a foundation for designing an intervention/interventions that may result in more patients achieving blood pressure control with maintained quality of life. Patients, who have well/not well controlled blood pressure, are to fill in questionnaires about their view on ability to perform self-care and their perceived quality of life. Individual interviews will also be made about for what reasons they do or do not change lifestyle as well as take their drugs to treat their hypertension. In focus group interviews the patients are to be asked about what they want and expect in the encounter with health care personnel, what other things outside the health care area would be helpful for the patient and how age, gender, cultural and psychosocial aspects affect the ability to achieve blood pressure control. The developed future interventions will be evaluated in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with hypertension since 9 months
* being able to read and speak Swedish

Exclusion Criteria:

-

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To preserve that the population is representative for an area in southern Sweden, patients are to be included consequtively through stratified sampling regarding age, gender and treatment at health centre or medical clinic at a hospital as well as geographically.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Self-care agency | through study completion, an average of 6 months
  Exercise of Self Care Agency (ESCA) instrument
Quality of life: SF-36 | through study completion, an average of 6 months
  Short Form Health Survey, 36 items
Individual interviews | through study completion, an average of 3 months
  Semistructured interviews
Focus-group interviews | through study completion, an average of 1 year
  Discussions in focus-groups

CONTACTS AND LOCATIONS:
Overall Officials: Lena-Karin Erlandsson, Principal Investigator — Department of Health Sciences
Locations (1):
- Department of Health Sciences, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Undecided